CLINICAL TRIAL: NCT04600804
Title: The Role of 18F-FDG-PET for Staging and Prognostication in Patients Enrolled in the Fondazione Italiana Linfomi (FIL) MCL0208 Trial
Brief Title: The Role of 18F-FDG-PET for Staging and Prognostication
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_MCL0208-PET
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Mantle Cell Lymphoma
Keywords: prognostic issues; PET review; MCL
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients registered in the MCL0208 trial: About 200 patients enrolled in the MCL0208 trial who performed the PET exams within the clinical trial and who consent to the present study: all PETs available at each center participating in this study will be collected and analyzed.
  In the clinical trial PET was optional at baseline (b-PET), before ASCT (i-PET) and after- ASCT (eot-PET). All the PETs available per patient will be collected and considered for analysis, both in the case PET are available at all the 3 time points above listed and in case of availability of PET at 1 or 2 time points only.

SUMMARY:
A retrospective, multicenter, non-interventional, imaging study ancillary to FIL_MCL0208 clinical trial (NCT02354313) in untreated adult patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
This is a retrospective, multicenter, non-interventional, imaging study devoted to patients diagnosed with MCL and enrolled in the MCL0208 international randomized, phase III clinical trial (NCT02354313).

The study is aimed at addressing a number of prognostic issues that still need to be clarified in MCL patients, by taking advantage of the PET performed within the MCL0208 trial and available for the analysis, and the clinical records and molecular data generated in the context of the trial.

In the clinical trial PET was optional at baseline (b-PET), before ASCT (i-PET) and after-ASCT (eot-PET), and none of the exams was used in the decisionmaking strategy. All the PETs available will be collected and considered for analysis. The study will not require additional treatment or procedures except those required for the MCL0208 trial. The participation of the patient to the MCL0208 trial is a pre-requisite to be involved in this study.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment of the patient in the MCL0208 clinical trial documented by the signature of the study informed consent;
* Patient's treatment in one of the centers that participated in the MCL0208 trial and that has joined the MCL0208-PET study as well;
* Evidence of signed informed consent for the MCL0208-PET study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 patients have been enrolled in the MCL0208 trial. We expect to analyze the PETs, clinical and biological data of about 200 patients enrolled in the MCL0208 trial who performed the PET exams within the clinical trial and who consent to the present study: all PETs available at each center participating in this study will be collected and analyzed.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity (proportion) and agreement (Cohen K) of PET results (performed in different time points) compared to the current standard (TC plus bone marrow biopsy). | 24 months
  To better define the role of PET for the staging of MCL patients at the time of diagnosis, for evaluation of response after induction treatment (pre-ASCT; i-PET) and post ASCT (eot-PET) in comparison to the current standards, namely computed axial tomography (CT) and bone marrow biopsy.
C-index, estimated comparing models adding or not PET parameters to standard prognostic factors in predicting PFS. | 24months
  To build a new prognostic model for PFS, including PET parameters, MIPI-b and biological data (e.g. MRD, GEP and mutational parameters).The achievement of these objectives could help to plan futures studies in order to improve the outcome of MCL patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mian, MD, Principal Investigator — Ematologia e Centro Trapianto Midollo Osseo, Ospedale di Bolzano, Italy
Locations (34):
- Italy (33):
  - Ematologia Ospedale Vito Fazzi, Lecce, Apulia
  - U.O.C Ematologia e Trapianto A.O. C. Panico, Tricase, Apulia
  - U.O.Ematologia Ospedale Guglielmo da Saliceto, Piacenza, Emilia-Romagna
  - Ematologia Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - U.O. di Ematologia Ospedale degli Infermi di Rimini, Rimini, Emilia-Romagna
  - S.O.C. Oncologia Medica A Centro Riferimento Oncologico, Aviano, Friuli Venezia Giulia
  - SOC Clinica Ematologica Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), Udine, Friuli Venezia Giulia
  - Ematologia Universitа Cattolica S. Cuore, Rome, Lazio
  - Ematologia Ospedale Policlinico San Martino S.S.R.L. - IRCCS per l Oncologia, Genoa, Liguria
  - U.O. Clinica Ematologica Ospedale Policlinico San Martino S.S.R.L. - IRCCS per l Oncologia, Genoa, Liguria
  - Ematologia ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Ematologia Ospedale Maggiore Policlinico - Fondazione IRCCS Ca Granda, Milan, Lombardy
  - SC Ematologia ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Ematologia ASST MONZA Ospedale S. Gerardo, Monza, Lombardy
  - Div. di Ematologia IRCCS Policlinico S. Matteo di Pavia, Pavia, Lombardy
  - U.O. Ematologia Istituto Clinico Humanitas, Rozzano, Lombardy
  - Unità Linfomi - Dipartimento Oncoematologia - Istituto Scientifico San Raffaele, Milan, Milan
  - S.C. Ematologia A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont
  - S.C. di Ematologia e Trapianto di Midollo Osseo A.O. S. Croce e Carle, Cuneo, Piedmont
  - SCDU Ematologia AOU Maggiore della Caritа di Novara, Novara, Piedmont
  - Ematologia Universitaria A.O.U. Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - S.C.Ematologia A.O.U. Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - SC Ematologia e CTMO Ospedale Businco, Cagliari, Sardinia
  - S.C. Ematologia Azienda Ospedali Riuniti Papardo-Piemonte, Messina, Sicily
  - Divisione di Ematologia A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo, Sicily
  - Divisione di Ematologia e T.M.O. - Ospedale Centrale di Bolzano, Bolzano, Trentino-Alto Adige
  - Unitа funzionale di Ematologia Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - S.C. Oncoematologia A.O. S. Maria di Terni, Terni, Umbria
  - S.C di Ematologia Ospedale Ca Foncello, Treviso, Veneto
  - U.O. Ematologia AOU Integrata di Verona, Verona, Veneto
  - Ematologia - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola
  - U.O. Ematologia - AOU Pisana, Pisa
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI), Trieste
- Instituto Português de Oncologia de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided